CLINICAL TRIAL: NCT04649866
Title: Vasculopathy and Remodeling of Coronary Arteries in FRDA Patients
Brief Title: Coronary Artery Disease in Patients With Friedreich's Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Principal Investigator, Stephen Y. Chan, Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY20070248
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich's ataxia; frataxin; cardiomyopathy
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies | interventions — Plethysmography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Endothelial dysfunction will be tested using Strain-gauge plethysmography to measure forearm blood flow during infusions of acetylcholine [ACh] and sodium nitroprusside [SNP]
  Interventions: Diagnostic Test: plethysmography
- Control group (Active Comparator): Endothelial dysfunction will be tested using Strain-gauge plethysmography to measure forearm blood flow during infusions of acetylcholine [ACh] and sodium nitroprusside [SNP]
  Interventions: Diagnostic Test: plethysmography

INTERVENTIONS:
Diagnostic Test: plethysmography — Forearm blood flow (FBF) measurements in both arms will be made using venous occlusion strain-gauge plethysmography prior to the initiation of any intra-arterial infusions. All FBF measurements will be expressed as mL/min per 100-1 mL forearm volume according to prior studies and the Whitney method.1, 2 Resting baseline FBF will be measured at least 30 minutes after venous and arterial catheter placement to ensure that blood flows in the cannulated arms are stabilized. We will measure FBF during the last 2 minutes of each infusion period. Infusions of individual vasoactive medications will occur over a 15-minute interval. There will be a 25-minute washout between vasoactive medications. Cumulative dose response curves will be constructed over 5-minute incremental infusions. We will proceed in the following order:
  * SNP 0.8, 1.6 and 3.2 mcg/min
  * ACh 7.5, 15 and 30 mcg/min
  * Normal saline

SUMMARY:
Friedreich's ataxia is a debilitating, inherited disease cause by mutations in a protein called frataxin (FXN). FXN is one of several proteins that controls the production of iron-sulfur clusters, molecules that are essential for energy production in our cells as well as repair of our genetic code embedded in DNA molecules. Friedreich's ataxia (FRDA) and deficiency of FXN results in a nerve disease affecting coordination and a condition called hypertrophic cardiomyopathy (HCM), marked by an abnormal thickening of the heart. Patients with HCM can then develop pulmonary hypertension (PH), a deadly condition of the blood vessels of the lung. While most of the research in FRDA has focused on nerves and heart muscle, alterations in blood vessels of the heart and lung may worsen disease in FRDA. But, the role of FXN in these blood vessels has never been defined.

Investigators pilot data suggest that Frataxin (FXN ) deficiency can control senescence and downstream function in various types of Endothelial cells (ECs), investigators hypothesize that Friedreich's Ataxia (FRDA) patients may demonstrate endothelial cells EC abnormalities throughout the vasculature potentially before overt cardiomyopathy develops.

DETAILED DESCRIPTION:
Procedure in details:

Investigators have extensive experience in the performance of forearm blood flow studies using strain gauge plethysmography in patient volunteers. Endothelial dysfunction will be tested according to methodologies employed in our blood flow laboratories for more than a decade. Strain-gauge plethysmography is used to measure forearm blood flow during infusions of acetylcholine [ACh], and sodium nitroprusside [SNP] . Intra-arterial infusions of acetylcholine to test endothelium-dependent blood flow. Acetylcholine acts on muscarinic receptors to increase intracellular calcium levels and activate endothelial nitic oxide (NO) synthase. SNP is an exogenous source of NO, to assess endothelium-independent vasodilatation.

Cumulative dose response curves will be constructed over 5-minute incremental infusions. Study doctor will proceed in the following order:

* SNP 0.8 1.6 and 3.2 mcg/min
* ACh 7.5 15 and 30 mcg/min
* Normal saline

Forearm blood flow (FBF) measurements in both arms will be made using venous occlusion strain-gauge plethysmography prior to the initiation of any intra-arterial infusions. Blood pressure and heart rate will be measured during the procedure through the ECG. All FBF measurements will be expressed as mL/min per 100-1 mL forearm volume according to prior studies and the Whitney method.1, 2 Resting baseline FBF will be measured at least 30 minutes after venous and arterial catheter placement to ensure that blood flows in the cannulated arms are stabilized. Study team will measure FBF during the last 2 minutes of each infusion period. Infusions of individual vasoactive medications will occur over a 15-minute interval. There will be a 25-minute washout between vasoactive medications. The ACh 30 mcg/min will run for a total of 10 minutes.

Test visit:

The study will consist of one visit. Research nurse will do the lab work once subject arrive (results will take about an hour), and if eligible study team will proceed with the research procedure.

All subjects scheduled for the visit will report to the CTRC on the morning of testing at 8:00 AM. The subject will be placed in a quiet room with a where he will meet with the study doctor and CRC. The study doctor will discuss with the subject the nature of the research study, the risks of study participation, and participants' rights as a research subject. Then will ask subject to sign consent form. After signing the consent form, the study doctor will perform screening procedure which include the following:

* Asking questions concerning all medications prescriptions and non-prescription medications (vitamins, herbal supplements, aspirin, etc.) that are presently taking. Study team will be recording all this information in the subject's research record.
* Obtain a medical history and physical examination conducted by the study doctor.
* Will record height, weight, and vital signs of the subject.
* Research nurse will draw blood for laboratory testing. These tests will be a complete blood count (a test to make sure that subject is not anemic, or have too few red blood cells), electrolytes (tests to check the chemistry levels), glucose, and clotting tests. These tests will be performed to evaluate the health of subjects' body during study participation. Approximately 1 1/2 tablespoons (22 mL) of blood will be collected for this sample.

All screening results will be reviewed by the study doctor prior to the procedure. Subject will be provided with any abnormal screening results so that he/she can follow up with their primary care doctor for further evaluation.

All results of these screening reports will be read by our study doctors before initiating the study, it is possible that after taking these tests subject may not be able to take part in this study. The total duration of this visit is approximately 3-4 hours.

Only 1 subject will be scheduled in the CTRC on any given testing day to meet appropriate clinical staffing requirements for the study.

The CTRC nurse will place a peripheral 20-22-gauge venous catheter in the subject's antecubital vein of the non-dominant forearm for the purpose of collecting initial blood draw that will be used for research. After confirmation and documentation of dual arterial perfusion of the hand by an Allen's test, Dr. Risbano (co-investigator), is a critical care physician and qualified in this critical care procedure with 19 years' experience of doing arterial lines, will place an 20-22 brachial artery catheter in the non-dominant arm for infusion and blood pressure monitoring. Any non-PI physician will be personally supervised by the PI for three cannulations before allowing independent cannulation. Prior to the brachial artery catheter placement 1% lidocaine will be administered by injection for local anesthesia. Brachial artery catheterization is required for the strain gauge approach to locally administer the drugs to the forearm arterial circulation, while limiting systemic effect. The intra-arterial catheter will be connected by a 3-way stopcock to a pressure transducer for blood pressure measurements and to an infusion pump. Blood Flow Measurements: Heart rate, cardiac rhythm, respirations, blood pressure, and oxygen saturation will be continuously monitored. Forearm blood flow measurements will be performed by means of strain gauge venous-occlusion plethysmography, using methodology employed by the PI at the Vascular Medicine Branch of NHLBI in many other studies. plethysmography cuff pressure is intermittent. A mercury-filled Silastic strain gauge is placed around the widest portion of the forearm, and connected to a plethysmograph calibrated to measure the percent change in volume. The plethysmograph is connected to a strip chart recorder for forearm blood flow measurements following inflation of a wrist cuff to suprasystolic pressure to exclude the hand circulation. The cuff is inflated for a duration of 8-10 seconds over a 15 second interval. A blood pressure cuff on the upper arm is inflated to 40 mmHg for 7 seconds with a rapid cuff inflator in order to occlude venous outflow, but not arterial inflow, into the forearm. This causes non invisible distention of the forearm at a rate proportionate to arterial inflow. Blood pressure will be recorded directly from the intraarterial catheter immediately after each series of flow measurements. The use of dual arm plethysmography will allow a direct comparison of the non-instrumented arm (as a control) with the instrumented arm (research procedure), and serial measurements collected every 15 seconds during the research process.

Upon completion of the research testing procedure, the study doctor will remove the venous and arterial catheters. A doctor will personally perform the decannulation procedure. The subject will be asked to remain in the supine position with the arm at or above heart level and to keep the arm still during the procedure. The doctor will ensure that all infusions are stopped and the stopcocks turned off to the patient. Any suture or tape used to secure the line will be removed using standard precautions. The cannula will then be removed and firm pressure held over the artery site with direct pressure of the thumb over sterile gauze for approximately 10 minutes at which time the doctor will check for any bleeding from the puncture site. If there is any bleeding, pressure will be held for an additional 10 minutes. Once there is no bleeding, a pressure dressing with Coban will be placed over the site. The subject will be instructed to remain in the supine position for an additional 10 minutes, and to remain in the study room for a 30-minute observation period. The arm will again be examined by the study physician prior to discharge of the subject at which time the doctor will instruct them regarding care of their arm and provide them with an instruction sheet.

Medical Record Information: Study team will request subject's authorization to access medical record information from their past, current and future medical record information related to their health condition to be recorded into the Research study. This information will be collected from Heart and Vascular Institute (HVI) records, hospital records and, if applicable, private physician records. Since heart failure symptoms/progression may change over time, and these changes may be important to this study result, future medical records will be collected indefinitely. The medical record information contained within the study database will be used for research related purposes for an indefinite time. Subjects medical record information may be reviewed to see if they were eligible for any ongoing or future research studies; if they were eligible, then study team may contact subjects.

Review of family history: For individuals who have a family history of FRDA, heart or lung disease, Study team may ask some basic information about other members of the family. Study team will not record in the Research study any identifiable information about individuals who have not signed consent to participate in this research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18
2. Has FRDA
3. Has recent clinical echocardiography data confirming normal cardiac function

Exclusion Criteria:

1. Patients younger than 18
2. Has abnormal cardiac function

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
vasomotor tone | 2-4 hours
  We will quantify vasomotor tone in regard to level of vasoconstriction and vasodilation at rest and in response to pharmacologic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chan, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Montefiore Hospital Clinical and Translational Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other individuals for future research and if shared will be shared without identifiers.
  Participant's medical record information contained within the Research study may be provided to secondary research investigators (i.e., research investigators who are not affiliated with the Comprehensive Pulmonary Hypertension Program at University of Pittsburgh). However, prior to its provision to any secondary investigators, the information shall be de-identified. The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will available starting 6 months after publication
Access Criteria: The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators